CLINICAL TRIAL: NCT00835887
Title: Relevance of Flavanols for Cardiovascular Function in End-Stage Renal Disease, a Phase 2 Study
Brief Title: Relevance of Flavanols for Cardiovascular Function in End-Stage Renal Disease
Acronym: ESRD
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: no patients recruited, responsible physician left clinic
Sponsor: RWTH Aachen University (Other)
Collaborators: Heinrich-Heine University, Duesseldorf (Other)
Responsible Party: Heinrich-Heine-University Düsseldorf, Department of Medicine, Divison of Cardiology, Pulmonology and Vascular Medicine
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ESRD-Study
Record Dates: First submitted 2009-02-03; First posted 2009-02-04 (Estimated); Last update posted 2015-09-23 (Estimated); Status verified 2015-09

CONDITIONS: End Stage Renal Disease
MeSH Terms: conditions — Kidney Failure, Chronic

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): Treatment with low dose flavanoids
  Interventions: Dietary Supplement: low and high dose flavanoids
- 2 (Experimental): Treatment with high dose flavanoids
  Interventions: Dietary Supplement: low and high dose flavanoids

INTERVENTIONS:
Dietary Supplement: low and high dose flavanoids — treatment with flavanoid-rich or flavanoid-low cacao twice daily

SUMMARY:
In this study, the acute and long-term effects of flavanols on vascular function in patients with ESRD will be investigated.

DETAILED DESCRIPTION:
In order to assess potential acute beneficial effects of flavanols in patients with ESRD, 10 patients undergoing dialysis will be recruited. Subjects will receive a cocoa drink with 16 mg, 250 mg, and 500 mg (in 100 mL water each) flavan-3-ols (40% epicatechine/catechine und 60% procyanidine), respectively, on three consecutively days. The functional/hemodynamic parameters (flowmediated dilation (FMD), venous-occlusion-plethysmography (VOP), blood pressure, heart rate), the biochemical marker of the circulating NO pool (nitrite, nitrate, RNOs), and the plasma levels of flavanols (epicatechine and catechine) will be determined before and after ingestion of the respective cocoadrink.

It is expected that flavanols dose-dependently improve vascular function and that this is associated with an increase in the circulating NO pool.

In order to assess long-term effects of flavanols on vascular function in patients with ESRD.

To characterize potential vascular long-term effects of flavanols in patients with ESRD, a placebo-controlled double-blinded randomized control study will be performed in 40 patients randomized in two groups. Patients will daily receive either a flavanol-poor cocoa drink or a flavanol-rich cocoa drink over a period of three months.

The flavanol-dosis that is necessary to affect vascular function will be assessed as described above. At the beginning of the study, after the first intake of the cocoa (in order to identify nonresponders) and monthly for a period of three months the vascular function will be assessed applying innovative imaging techniques to the brachial artery to assess endothelium-dependent regulation of physicomechanical properties and vascular tone and thus blood flow at the level of the macrocirculation. In parallel new techniques will be applied to assess perfusion at the level of the microcirculation. In particular, measurement of flow-mediated dilation, intima-media-thickness,compliance and stiffness indices will be performed in the macrocirculation of the brachial artery.

Considering the microcirculation, new diagnostic approaches such as Laser-Doppler Flow and peripheral arterial tonometry next to diagnostic approaches such as the venous occlusive plethysmography will be performed. Moreover, the circulating NO pool, markers of inflammation and of oxidative stress, the uremic toxin pcresol and the plasma levels of flavanols will be determined. The exams after month 1, 2, and 3 will be performed in the morning before intake of the cocoa drink. In order to examine potential sustained effects, an additional examination day will take place after 4 month (one month after stopping the flavanol-intake). It is expected that the flavanol-rich cocoa will improve vascular function, which is associated with an increase in the circulating NO-pool and a decrease in inflammatory markers and the marker for oxidative stress.

ELIGIBILITY:
Inclusion Criteria:

* patients with end stage renal disease

Exclusion Criteria:

* person under 18 years of age
* participation in another study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)

PRIMARY OUTCOMES:
Vascular function | before treatment, directly after treatment and 3, resp. 4 months afterwards

CONTACTS AND LOCATIONS:
Locations (1):
- Düsseldorf University Hospital, Düsseldorf, Germany